CLINICAL TRIAL: NCT01258413
Title: Laparoscopic vs Abdominal Radical Hysterectomy With Pelvic Lymphadenectomy in Patients With Early Cervical Cancer: A Randomized Clinical Trial
Brief Title: Laparoscopic vs Abdominal Radical Hysterectomy In Patients With Early Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Dr. Leo Franscisco Limberger, Hospital Nossa Senhora da Conceição
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPGHC: 65/99
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-11

CONDITIONS: Cervical Cancer; Postoperative Pain
Keywords: Cervical Cancer; Radical hysterectomy, Laparoscopic; Overall survival; Disease-free five-years survival
MeSH Terms: conditions — Uterine Cervical Neoplasms; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Radical Hysterectomy (Experimental): uterus, upper 1-2cm of vagina , parametrial tissue and uterosacral ligament are removed + pelvic lymphadenectomy
  Interventions: Procedure: Laparoscopic Radical Hysterectomy + pelvic lymphadenectomy
- Abdominal radical hysterectomy (Active Comparator): uterus, upper 1-2cm of vagina , parametrial tissue and uterosacral ligament are removed + pelvic lymphadenectomy
  Interventions: Procedure: Abdominal radical hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic Radical Hysterectomy + pelvic lymphadenectomy — uterus, upper 1-2cm of vagina , parametrial tissue and uterosacral ligament + pelvic lymphadenectomy are removed by laparoscopic approach
  Arms: Laparoscopic Radical Hysterectomy
Procedure: Abdominal radical hysterectomy — uterus, upper 1-2cm of vagina , parametrial tissue and uterosacral ligament + pelvic lymphadenectomy are removed by abdominal approach
  Arms: Abdominal radical hysterectomy

SUMMARY:
The purpose of this study is to determine whether laparoscopic radical hysterectomy for early cervical cancer will has decreased postoperative pain intensity compared to abdominal radical hysterectomy with similar postoperative complications and survival rates.

DETAILED DESCRIPTION:
Background: Radical hysterectomy with pelvic lymphadenectomy is one of the FIGO (International Federation of Gynecology and Obstetrics) recommended treatments for early cervical cancer. The objective of this study was to compare radical hysterectomy by laparoscopic approach and open radical hysterectomy in a single center randomized clinical trial. Nevertheless, there are no finished randomized controlled trials comparing laparoscopic radical hysterectomy and abdominal radical hysterectomy although there is an ongoing trial.

Methods: Were enrolled 30 IA2 with lymph vascular space invasion and IB cervical cancer patients. Postoperative pain intensity was defined as primary endpoint and pain intensity was measured by a 10-point numeric rating scale. Secondary outcomes were: intraoperative and other postoperative outcomes, histopathological outcomes and 5-year follow-up. Data analysis is being done at this moment

ELIGIBILITY:
Inclusion Criteria:

* Women of 18 years or older referred to our service with histologically confirmed primary squamous, adenocarcinoma or adenosquamous cervical cancer diagnosed by biopsy or cervical conization, clinically FIGO (International Federation of Gynecologic and Obstetrics) staged IA2 with lymph vascular invasion, IB and II A.

Exclusion Criteria:

* Patients with clinically advanced disease (IIB-IV), previous pelvic or abdominal radiotherapy, pregnancy, clinical diseases that would preclude one or both surgical approaches.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-11; Primary Completion 2004-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
postoperative pain measured by a 10 point numeric rating scale | around one week
  The primary outcome is postoperative pain as measured by a 10-point numeric rating scale (NRS) during the postoperative period. Pain was assessed every six hours by nursing staff during a patient's usual postoperative care. The nursing staff was not aware of the study objective.

SECONDARY OUTCOMES:
Intraoperative, perioperative and postoperative complication | 30 days or five years
  1 Intraoperative outcomes included the following: operative time (minutes), injuries to the ureter, bladder, bowel or vessels and anaesthesia complications requiring blood transfusion.
  2. Early (< 30 days) or late postoperative events and findings during the hospital stay or after included the following: hospital stay duration (days), complications. Surgical or clinical findings that could be attributable to the treatment in five years of follow up 74 Clinical or surgical findings that could be attributable to the treatment or the disease at five years of follow-up.
Surgicopathological outcomes | postoperatively
  outcomes included the following: histological type, surgical margins, lymph node status and lymph node number, all assessed by pathologists with expertise in gynaecologic oncology. In addition, parametrial and vaginal cuff width (centimetres) was assessed by the first surgeon in the operating room, before tissue processing.
Overall survival and disease-free survival | five years
  Clinical status in the last visit recorded; Date and location of the first recurrence or metastasis. Time frame: five years from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Leo F Limberger, M.D., Principal Investigator — Hospital Nossa Senhora da Conceição
Locations (1):
- Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Campos LS, Limberger LF, Stein AT, Kalil AN. Postoperative pain and perioperative outcomes after laparoscopic radical hysterectomy and abdominal radical hysterectomy in patients with early cervical cancer: a randomised controlled trial. Trials. 2013 Sep 12;14:293. doi: 10.1186/1745-6215-14-293. PMID 24028441